CLINICAL TRIAL: NCT02261142
Title: Evaluation of Efficacy and Cost-effectiveness of Spasticity Treatment With Multifocal Transcutaneous Electrical Stimulation, Through a Garment With built-in Electrodes in Combination With Training.
Brief Title: Efficacy and Cost-effectiveness of Spasticity Treatment With Multifocal TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: University of Borås (Unknown); University Hospital, Linkoeping (Other); Sodra Alvsborgs Hospital (Other)
Responsible Party: Principal Investigator, Per Ertzgaard, M.D., Linkoeping University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIU-ED2013
Record Dates: First submitted 2014-10-01; First posted 2014-10-10 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Spasticity; Stroke; Cerebral Palsy
MeSH Terms: conditions — Muscle Spasticity; Stroke; Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifocal TENS (Experimental): Multifocal TENS given in the garment Mollii® (Elektrodress) 1 hour every second day together with individualized training exercises. The steering unit counts down 60 minutes visible for the patient
  Interventions: Device: Multifocal TENS garment (Mollii®)
- Sham treatment (Sham Comparator): Use of the garment Mollii® (Elektrodress) but without the electrical stimulation combined with the individualized training exercises. The steering unit counts down 60 minutes visible for the patient
  Interventions: Device: Multifocal TENS garment (Mollii®)

INTERVENTIONS:
Device: Multifocal TENS garment (Mollii®) — Multifocal transcutaneous electrical stimulation incorporated into a whole-body garment in combination with training
  Other Names: Mollii®; Elektrodress; Swedish patent:SE534365.C2

SUMMARY:
Spasticity is a common consequence of injury to the central nervous system and can be a major problem in motor function and everyday activities. A method for treating spasticity that applies low-amplitude electrical stimulation through a garment with built-in electrodes, Mollii® (Elektrodress), has been developed. The garment is to be used in combination with individualized training and the stimulation is mainly given to antagonists of spastic muscles.

The general objective of this study is to evaluate the efficacy of and costs associated with the Mollii® treatment of spasticity due to stroke or cerebral palsy.

Primary objectives are;

* to study whether treatment with the Mollii® improves function and activity
* to evaluate the cost-effectiveness of the treatment, from both a health-care perspective and a societal perspective.

Secondary objectives are;

* to study whether there are differences in treatment effect between the stroke and the Cerebral Palsy groups in a subgroup-analysis
* to assess compliance with treatment
* to report any adverse effects.

DETAILED DESCRIPTION:
This study is designed as a double-blinded, randomized, cross-over trial (RCT). This part of the study takes 12 weeks (6 weeks of active treatment and 6 weeks of non-active treatment) and is followed by a wash-out period of 6 weeks. An uncontrolled,open phase starts after week 18, where patients are followed one year after inclusion.

30 participants with spasticity due to Stroke and Cerebral Palsy will be included.

Two centers are recruiting participants and are collecting data.

Outcome measures are chosen to reflect the different dimensions in the International Classification of Functioning, Disability and Health (ICF) and patient reported outcome measures (PROM).

ELIGIBILITY:
Inclusion Criteria:

* Spasticity due to stroke or Cerebral Palsy
* Have some preserved walking ability, with or without walking aids
* Be able to understand the treatment and instruments/interviews used
* For stroke participants, two years should have elapsed since their injury/insult

Exclusion Criteria:

* Electronic devices
* Ventriculoperitoneal shunt
* Arrhythmia
* Hearth infarction or unstable angina pectoris
* Symptomatic hyper- or hypotonia
* Cancer under treatment
* Unstable psychiatric disease
* Lung disease, affecting daily life
* Unstable epileptic disease
* Orthopedic surgery last year
* Obesity with BMI > 35
* Infectious disease with longstanding treatment
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Goal attainment scaling (GAS) | 12 weeks
  1 to 3 goals are defined and evaluated using the original GAS scale by Kiresuk
Arm-hand ability (ARAT + WMFT tasks 1&2) | 12 weeks
  Action Research Arm Test (ARAT)measuring grasp, grip, pinch and gross movement and this is complemented by Wolf Motor Function Test (WMFT) tasks 1 and 2 measuring active shoulder abduction
Mobility | 12 weeks
  10 meter walking test, divided into comfortable gait test (CGT) and fast gait test (FGT). Outcome is velocity, cadence and stride length.
  Timed Up & Go (TUG)

SECONDARY OUTCOMES:
Health related Quality of Life/QALY | Baseline, week 6, 12, 18, 52
  SF-36 and EQ-VAS
Self reported pain and spasticity | Baseline, week 6, 12, 18, 52
  Numeric rating scale (NRS)
Muscle hypertonicity (Spasticity) | Baseline, week 6, 12, 18, 52
  Modified Ashworth scale (0-5)
Range of Motion | Baseline, week 6, 12, 18, 52
  Goniometer
Costs | Baseline, week 6, 12, 18, 52
  Costs directly related to intervention Baseline, week 6, 12, 18 Costs from a societal perspective at baseline and week 52
Goal Attainment Scaling (GAS) | 52 weeks
  1 to 3 goals are defined and evaluated using the original GAS scale by Kiresuk
Arm-hand ability (ARAT + WMFT tasks 1&2) | 52 weeks
  Action Research Arm Test (ARAT)measuring grasp, grip, pinch and gross movement and this is complemented by Wolf Motor Function Test (WMFT) tasks 1 and 2 measuring active shoulder abduction
Mobility | 52 weeks
  10 meter walking test, divided into comfortable gait test (CGT) and fast gait test (FGT). Outcome is velocity, cadence and stride length.
  Timed Up & Go (TUG)